CLINICAL TRIAL: NCT02574780
Title: Lymphedema Treatment of Post-surgical Upper Limb of Breast Cancer Through Muscle Strengthening Associated With Complex Physical Therapy
Brief Title: Lymphedema Upper Limb of Breast Cancer Through Muscle Strengthening Associated With Complex Physical Therapy
Acronym: LTP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Gil Facina, Doctor clinical, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUSaoPaulo,PT 1
Record Dates: First submitted 2015-10-09; First posted 2015-10-14 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Lymphedema
Keywords: lymphedema; complex physical therapy; muscle strength
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Grupo I TFC (Experimental): Women with lymphedema , perform complex physical therapy with manual lymphatic drainage, compression bandaging and exercises linfomiocinéticos.
  Interventions: Other: complex physical therapy; Other: Evaluate treatment of lymphedema, with in the quality of life and depression
- Grupo II TFC X PFM (Experimental): Standard treatment for lymphedema perform complex physical therapy associated with a muscular strength protocol.Muscle-building arm with load
  Interventions: Other: complex physical therapy; Other: Evaluate treatment of lymphedema, with in the quality of life and depression

INTERVENTIONS:
Other: complex physical therapy — Compare the standard treatment of lymphedema, by complex physical therapy versus TFC associated with the upper limbs strengthening exercises.
Other: Evaluate treatment of lymphedema, with in the quality of life and depression — evaluate through the questionnaires fatigue and quality of life of patients with lymphedema (FACT- F and Inventory BECK)

SUMMARY:
The stage and lymphedema size can be detrimental to the quality of life and health of women, because the increase in circumference and member of the weight causes limitations in activities. Previous studies have shown that patients with lymphedema should not perform high intensity exercises, these exercises would cause the increase of lymphedema. Already, in current studies show that muscle strength exercises when properly applied, with controlled intensity and time, can help to reduce lymphedema. Thus, the main objective of this study is to compare the standard treatment of lymphedema through complex physical therapy versus the application of strengthening exercises for upper limbs together with complex physical therapy. The study design is a randomized controlled clinical trial. Participate in the study 50 patients, who will be allocated into two groups, group 1 (n = 25): Complex Physical Therapy; Group 2 (n = 25): Complex physical therapy in an exercise protocol, which will receive treatment twice a week for eight weeks. All patients will receive treatment and will be informed of the free and informed consent form at the beginning of the research. They will be met: the report cards, dynamometer testing and filling out questionnaires at the beginning and end of the study.

DETAILED DESCRIPTION:
This study will be conducted in Onco Mastology clinic of the Department of Mastology the Department of Gynecology, Federal University of São Paulo (UNIFESP) - Paulista School of Medicine (EPM), in which patients will be recruited, selected and informed about the study objectives , its relevance, activities to be developed and the possibility of improvement and remedy your questions and concerns about the disease.The study design is a randomized controlled clinical trial. To define the treatment, 50 patients are allocated to two groups, group 1 (n = 25) Group 2 (n = 25) that receive treatment twice a week for eight weeks. Physical examination will be performed, completing the consent form, evaluation form, and questionnaires. Group 1 standard treatment : 25 women with lymphedema , perform complex physical therapy with manual lymphatic drainage, compression bandaging and exercises linfomiocinéticos . Treatment was given twice a week , 8 consecutive weeks , 6 sessions.Group 2 standard treatment + muscle strength : 25 women with lymphedema , perform complex physical therapy, manual lymphatic drainage, compression bandaging and linfomiocinéticos exercises and strengthening exercises with load.Treatment was given twice a week , 8 consecutive weeks , 16 sessions.

ELIGIBILITY:
Inclusion Criteria:

* With lymphedema resulting from postoperative unilateral breast cancer
* difference in circumference between the upper limbs

Exclusion Criteria:

* Patients with bilateral breast cancer
* Grade IV lymphoedema called elephantiasis
* renal dysfunction
* treatment involving the reduction of lymphedema in the last three months; acute inflammation ; deep vein thrombosis ; heart disease; skin infections and disease locoregional or distant active base.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Result of complex physical therapy associated with muscle strength protocol | two years
  Brawn average difference between the upper limbs with and without lymphedema.

CONTACTS AND LOCATIONS:
Overall Officials: Gil Facina, Principal Investigator — BRazil:Research committee - Recruting
Locations (1):
- Brazil Federal University São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No